CLINICAL TRIAL: NCT02527018
Title: A Comparison of B Type Natriuretic Peptide Levels and Hemodynamics Using the Nexfin Device in Healthy Pregnant and Preeclamptic Women - A Pilot Study
Brief Title: A Comparison of BNP Levels Using the Nexfin Device in Healthy Pregnant and Preeclamptic Women
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Afshan B. Hameed, M.D., Associate Professor of Clinical OBGYN / Medical Director Obstetrical Services for OBGYN, University of California, Irvine
Other Study IDs: 2014-1232
Record Dates: First submitted 2015-07-29; First posted 2015-08-18 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Preeclampsia; Maternal; Hypertension; Pregnancy
Keywords: OBGYN; Nexfin; Hypertensive; Hemodynamic
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Sphygmomanometers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Subjects: Measurement of hemodynamic levels (BNP) of healthly term subjects using the Nexfin sphygmomanometer device.
  Interventions: Device: Sphygmomanometer
- Preeclamptic Subjects: Measurement of hemodynamic levels (BNP) of preeclamptic subjects using Nexfin sphygmomanometer device.
  Interventions: Device: Sphygmomanometer

INTERVENTIONS:
Device: Sphygmomanometer — Non-invasive reliable method of continuous measuring arterial blood pressure in pregnant women. Nextfin provides continuous blood pressure, heart rate, cardiac output, stroke volume, systemic vascular resistance and left ventricular contractility indices.
  Other Names: Nextfin

SUMMARY:
Primary Endpoint: Quantify the hemodynamic changes in preeclampsia using the non-invasive Nexfin device.

Secondary Endpoint: Determine if measurable hemodynamic changes are statistically correlated with B-type natriuretic peptide (BNP) levels.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy including preeclampsia are the leading cause of pregnancy related mortality in the United States. Timely and appropriate management of hypertensive disorders of pregnancy is critical to prevent complications such as kidney failure, HELLP syndrome, disseminated intravascular coagulation, placental abruption, intrauterine fetal demise, intracranial bleed, coma and death. (HELLP syndrome is a group of symptoms that occur inpregnant women who have: H -- hemolysis (the breakdown of red blood cells); EL -- elevated liver enzymes; LP -- low platelet count.) Hypertensive disorders of pregnancy include gestational hypertension (HTN), chronic HTN, preeclampsia and preexisting HTN with superimposed preeclampsia.

Hypertensive disorders may also lead to significant maternal and/or fetal morbidity. Based on the severity of the disease process and gestational age of the fetus, decision needs to be made whether to proceed with immediate delivery or continue expectant management. Meanwhile, maintenance of optimal blood pressure, blood volume, and cardiac output are recommended to preserve placental perfusion and to prevent unfavorable maternal and/or fetal outcomes.

Previous studies have demonstrated blood flow differences in pregnancies complicated by preeclampsia vs. healthy pregnant women evidenced by decreased arterial compliance, increased systemic vascular resistance and after load, and changes in blood volume and cardiac output. Additionally, various serum markers have been tried to identify women with preeclampsia. B-Type natriuretic peptide (BNP) has been consistently shown to be elevated in preeclampsia, and serves as a marker of heart function and intra vascular volume status.

Continuous hemodynamic monitoring may play a crucial role in timely management of these patients with severe disease due to the dynamic nature of the disease process. Existing methods are not preferred in pregnancy due to their invasive nature, and there is lack of validated non-invasive means to provide real time information on various hemodynamic parameters including cardiac output in these critically ill pregnant women.

Among new cardiac monitoring devices, the Nexfin device (BMEYE, Amsterdam, Netherlands) has recently been introduced. Nexfin device is a device approved by the Food and Drug Administration (FDA) as a non-invasive reliable method of continuous measuring arterial blood pressure in pregnant women. However there are no preliminary data on preeclamptic patients using this device. The standard of care is to use a sphygmomanometer for blood pressure monitoring. Additionally there are no studies comparing the hemodynamics of healthy and preeclamptic women using Nexfin device. Nexfin is thought to be superior over other available non-invasive methods as it is a safe and a considerably accurate method. Nexfin provides continuous blood pressure, heart rate, cardiac output, stroke volume, systemic vascular resistance and left ventricular contractility indices.

The study aims to determine if the non-invasive Nexfin device can be used to reliably distinguish hemodynamics in preeclamptic vs. healthy pregnant women with singleton pregnancies along with use of BNP levels. Investigators aim to recruit 33 healthy controls and 33 subjects diagnosed with preeclampsia (mild and severe). Subject's systolic and diastolic blood pressures will be measured using both the Nexfin device and a standard sphygmomanometer (blood pressure meter). Additionally hemodynamic measure such as: heart rate, cardiac output, stroke volume, systemic vascular resistance, and left ventricular contractility will be recorded using the Nexfin device. Investigators will perform a blood draw to measure BNP levels as an additional assessment of the hemodynamic changes in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged (x> or =18) with or without preeclampsia.
* Subjects with preeclampsia must have either mild or severe preeclampsia
* Healthy subjects should be normotensive
* Gestational age between 28 weeks to 40 0/7 weeks

Exclusion Criteria:

* Pregnant women aged (x<18)
* Pregnant women with multiple gestations
* Diagnosis of cardiac disease
* Diagnosis of vascular disease
* Diagnosis of end stage renal disease
* Subjects in active labor
* Diagnosis of Systemic Lupus Erythematosus or any other autoimmune disease
* Fetus' known to have age abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 33 healthy controls and 33 subjects diagnosed with preeclampsia (mild and severe).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Composite Hemodynamic Preeclamptic Changes | One hospital visit (duration 30 minutes).
  Composite Changes are defined by volume overload (mL), higher B-type natriuretic peptide levels pg/mL, higher blood pressure or cardiac output (mm / Hg).

SECONDARY OUTCOMES:
Composite Statistical Correlation For Normotensive and Preeclamptic Subjects | One hospital visit (duration 30 minutes).
  Composite Statistical Correlation are defined by systolic (SBP) and diastolic (DBP) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Afshan Hameed, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Department of OBGYN, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No